CLINICAL TRIAL: NCT06235515
Title: Does Adding Virtual Reality Therapy to Conventional Physical Therapy Improve Clinical Outcomes in Individuals With Chronic Neck Pain?
Brief Title: Additional Benefits of Virtual Reality Therapy for Individuals With Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Nazife Kapan, Asst. Prof., Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AEÜ-NK-SG
Record Dates: First submitted 2024-01-08; First posted 2024-02-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Neck Pain; Virtual Reality; Rehabilitation
MeSH Terms: conditions — Neck Pain | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group I (Experimental): conventional treatment As conventional treatment, patients will receive 20 minutes of hotpack and 20 minutes of TENS, 5 sessions a week for a total of 15 sessions for 3 weeks. Additionally, patients will be given cervical isometric exercises as a home exercise program.
  Interventions: Other: rehabilitation program
- group II (Experimental): conventional treatment and virtual reality As conventional treatment, patients will receive 20 minutes of hotpack and 20 minutes of TENS, 5 sessions a week for a total of 15 sessions for 3 weeks. Additionally, patients will be given cervical isometric exercises as a home exercise program.
  In addition to conventional treatment, virtual reality treatment will allow patients to play games in which they can perform neck movements in all directions for 30 minutes a day, 5 sessions a week for 3 weeks..
  Interventions: Other: rehabilitation program; Other: virtual reality

INTERVENTIONS:
Other: rehabilitation program — conventional treatment (hotpack and TENS and exercise)
Other: virtual reality — virtual reality treatment
  Arms: group II

SUMMARY:
This study aimed to investigate the effect of adding virtual reality therapy to conventional treatment in patients with chronic neck pain on pain, neck disability index, kinesiophobia, insomnia severity questionnaire, hospital anxiety depression scale, cervical range of motion and pressure pain threshold.

DETAILED DESCRIPTION:
Neck pain is a disease that affects individuals and society worldwide. Between 50% and 85% of the general population experiences neck pain at some point in their lives, and every person who experiences neck pain is likely to experience pain again after 1-5 years. Neck pain is considered chronic if it lasts more than 3 months. Passive and active physical therapy approaches play a very important role in the treatment of neck pain. With the rapid development of technology, new developments such as virtual reality have begun to be used in the treatment of chronic neck pain.

Virtual reality (VR) is a term describing innovative, real-time, computer-based technologies that play an increasing role for many patient groups in the field of physical medicine and rehabilitation. Virtual reality has been shown to be effective in reducing pain and discomfort in patients with different types of chronic pain. Motivation and interaction are the main practical benefits of virtual reality training, especially in video game-based therapy approaches, unlike traditional rehabilitation. Patients play the therapeutic game over and over again to achieve a better score without getting bored. Feedback, an important component of motor learning, is a prominent feature in virtual environments.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 who signed the informed consent form
* Those with existing neck pain
* Those whose neck pain continues for at least 12 weeks

Exclusion Criteria:

* Previous cervical surgery
* Having received FTR from the cervical region in the last 6 months
* Having had a spinal fracture
* History of malignancy
* Those with pacemakers
* Those with rheumatological, vestibular and neurological diseases
* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2024-09-16 (Actual)

PRIMARY OUTCOMES:
Visual Anolog Scale | Before treatment and three weeks
  It is a pain rating scale with numbers 0 and 10. Here 0 means 'no pain' and 10 means 'unbearable pain'. The participant will rate the pain according to the scale. Patients' night, rest and activity pain will be evaluated separately.
Neck Disability Index | Before treatment and three weeks
  It is the most widely used scale for cervical dysfunction and pain. It is also a unidimensional measurement used to determine the patient's perceived level of disability due to neck pain. It is a personal questionnaire consisting of 10 items regarding daily living activities. Each section is scored from 0 (no disability) to 5 (complete disability). The total score ranges from 0 (no injury) to 50 (total injury).
Range of Motion | Before treatment and three weeks
  Cervical range of motion, flexion, extension, right-left lateral flexion and right-left rotations will be measured and recorded using a goniometer. Normal joint ranges of motion; Flexion was determined as 50 degrees, extension as 70 degrees, lateral flexion as 45 degrees and rotation as 80 degrees.

SECONDARY OUTCOMES:
Tampa Kinesiophobia Scale | Before treatment and three weeks
  It consists of 17 questions designed to measure fear of movement. A 4-point Likert scoring (1: strongly disagree, 2: disagree, 3: agree, 4: completely agree) is used. Total score varies between 17-68. It is concluded that the higher the person scores on the scale, the higher the fear of movement.
Insomnia Severity Index | Before treatment and three weeks
  This scale, developed to determine the degree of insomnia symptoms, can be used in normal population screening and clinical evaluation of insomnia. It is a five-point Likert type scale consisting of seven items. 0-7 points indicate insignificant insomnia, 8-14 indicates clinically subthreshold insomnia, 15-21 indicates moderate insomnia, and 22-28 indicates severe insomnia.
Hospital Anxiety Depression Scale | Before treatment and three weeks
  This scale was used to determine anxiety and depression symptomatology. The scale consists of a total of 14 items, 7 items assessing depression and 7 items assessing anxiety. By summing the subscale scores, 0-21 points can be obtained from each of the depression and anxiety scales. 0-7 points; no depression or anxiety disorder, 8-10 points; mild depression or anxiety disorder, 11-14 points; moderate, 15-21 points; indicates severe disorder.
Pressure Pain Threshold | Before treatment and three weeks
  A pressure algometer (Baseline dolorimeter-66 pound sensitivity- with circular probe) will be used to evaluate the pressure pain threshold. Pain pressure thresholds will be measured from both the right and left upper trapezius and the right-left C1/2 and C5/6 articular pilar level. Before measurements are taken at these points, the pressure pain threshold measurement will be displayed on the patient's hand in order to familiarize the patient with the procedure. Participants will be told to say 'stop' when the feeling changes from pressure to pain. Three measurements will be made at each point with a 1 cm diameter probe and a maximum pressure of up to 60 N will be applied at a speed of approximately 3 N/s. A 30-second rest period will be left between each measurement and the average of the measurements will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran University, Kırşehir, Turkey (Türkiye)

REFERENCES:
- [Background] Haldeman S, Carroll L, Cassidy JD. Findings from the bone and joint decade 2000 to 2010 task force on neck pain and its associated disorders. J Occup Environ Med. 2010 Apr;52(4):424-7. doi: 10.1097/JOM.0b013e3181d44f3b. PMID 20357682
- [Background] Vernon HT, Humphreys BK, Hagino CA. A systematic review of conservative treatments for acute neck pain not due to whiplash. J Manipulative Physiol Ther. 2005 Jul-Aug;28(6):443-8. doi: 10.1016/j.jmpt.2005.06.011. PMID 16096044
- [Background] Ahern MM, Dean LV, Stoddard CC, Agrawal A, Kim K, Cook CE, Narciso Garcia A. The Effectiveness of Virtual Reality in Patients With Spinal Pain: A Systematic Review and Meta-Analysis. Pain Pract. 2020 Jul;20(6):656-675. doi: 10.1111/papr.12885. Epub 2020 May 21. PMID 32196892
- [Background] Adamovich SV, Fluet GG, Tunik E, Merians AS. Sensorimotor training in virtual reality: a review. NeuroRehabilitation. 2009;25(1):29-44. doi: 10.3233/NRE-2009-0497. PMID 19713617
- [Background] Burdea GC. Virtual rehabilitation--benefits and challenges. Methods Inf Med. 2003;42(5):519-23. PMID 14654886
- [Background] Holden MK. Virtual environments for motor rehabilitation: review. Cyberpsychol Behav. 2005 Jun;8(3):187-211; discussion 212-9. doi: 10.1089/cpb.2005.8.187. PMID 15971970